CLINICAL TRIAL: NCT01844700
Title: 1/2-MC4R Genotype and Pediatric Antipsychotic Drug- Induced Weight Gain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: very slow recruitment, no sufficient results
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Anil K. Malhotra, Director, Psychiatric Research, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 12-403A
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: High Risk MC4R Genotype; Low Risk MC4R Genotype; One Week or Less Antipsychotic Lifetime Exposure
Keywords: MC4R genotype; antipsychotic induced weight gain; pediatric population
MeSH Terms: interventions — ziprasidone; Aripiprazole; Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ziprasidone (Active Comparator): (20-160mg/d, bid) for 12 weeks
  Interventions: Drug: Ziprasidone
- Aripiprazole, quetiapine, risperidone (Active Comparator): Aripiprazole (2-30mg/d), Quetiapine (25-800mg/d) or Risperidone (0.1-8mg/d) for 12 weeks
  Interventions: Drug: aripiprazole, quetiapine, or risperidone

INTERVENTIONS:
Drug: Ziprasidone — random assignment to ZIP (20-160mg/d, bid dosing)
  Other Names: Geodon
  Arms: Ziprasidone
Drug: aripiprazole, quetiapine, or risperidone — random assignement to Usual Care antipsychotic UC antipsychotic (aripiprazole 2-30mg/d, quetiapine 25-800mg/d or risperidone 0.1-8mg/d)
  Other Names: Abilify, Seroquel, Risperdal
  Arms: Aripiprazole, quetiapine, risperidone

SUMMARY:
We will conduct a 12-week, randomized open label study, comparing usual care (UC) antipsychotic treatment (aripiprazole, quetiapine, risperidone) with ziprasidone (ZIP) in children and adolescents aged 13-18 years old. Patients will have 10 days or less lifetime antipsychotic exposure and be in clinical need for antipsychotic treatment for a pediatric psychiatric disorder with FDA indication for antipsychotic use, i.e., bipolar mania, schizophrenia-spectrum disorders, and irritability associated with autistic disorder. In addition, we will also include youth fulfilling research diagnostic criteria for severe mood dysregulation (SMD). Randomization will be stratified by high vs. low genetic risk for antipsychotic-induced weight gain based on MC4R genotype and the primary outcome will be weight change from baseline to endpoint between ZIP and UC antipsychotic treatment in each of the two genotype groups. As detailed below, other metabolic and cardiac safety parameters will also be measured and compared across treatments in each of the genotype groups.

ELIGIBILITY:
Inclusion Criteria:

* age 13-18 years
* English-speaking
* DSM diagnoses that have an FDA indication for SGA use for at least one agent in the respective pediatric or adult age group. Specifically, primary DSM-IV diagnosis of early-onset schizophrenia spectrum disorders; bipolar I disorder mania (and BP-NOS); irritability associated with autism spectrum disorder, as well as severe mood dysregulation (SMD) according to Leibenluft et al. (2011) with an ABC-irritability score of >/=18 Sexually active girls must agree to use two effective forms of birth control or be abstinent
* Participant has a primary caretaker who has known the child well for at least 6 months before study entry Primary caretaker is able to participate in study appointments
* Ability of child to participate in all aspects of the protocol per investigator clinical judgment.

Exclusion Criteria:

* Major neurological or medical illnesses that affect weight (e.g., unstable thyroid disease), require a prohibited systemic medication (e.g., diabetes mellitus [insulin], chronic renal failure [steroids); Fasting glucose > 125 mg/dL on 2 occasions during screening
* Any medication (other than currently prescribed psychotropic medications) that would significantly alter weight
* Antidepressants not allowed for at least 2 weeks in BP-I or BP-NOS patients
* DSM-IV diagnosis of anorexia or bulimia nervosa
* DSM-IV diagnosis of Substance Dependence disorder (other than tobacco dependence) within the past month
* Initial urine toxicology screen and follow-up screen indicate ongoing use of illicit substance
* Hypersensitivity to ZIP or UC antipsychotics
* Pregnant, breast feeding or unwilling to comply with contraceptive requirements
* Screening or baseline QTc > 450 msec
* IQ < 55
* Significant risk for dangerousness to self or to others
* Ongoing or previously undisclosed child abuse requiring new department of social service intervention.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Zucker Hillside Hospital, Psychiatry Research, Glen Oaks, New York, United States

REFERENCES:
- [Background] Allison DB, Mentore JL, Heo M, Chandler LP, Cappelleri JC, Infante MC, Weiden PJ. Antipsychotic-induced weight gain: a comprehensive research synthesis. Am J Psychiatry. 1999 Nov;156(11):1686-96. doi: 10.1176/ajp.156.11.1686. PMID 10553730
- [Background] Axelson D, Birmaher B, Strober M, Gill MK, Valeri S, Chiappetta L, Ryan N, Leonard H, Hunt J, Iyengar S, Bridge J, Keller M. Phenomenology of children and adolescents with bipolar spectrum disorders. Arch Gen Psychiatry. 2006 Oct;63(10):1139-48. doi: 10.1001/archpsyc.63.10.1139. PMID 17015816
- [Background] Basile VS, Masellis M, McIntyre RS, Meltzer HY, Lieberman JA, Kennedy JL. Genetic dissection of atypical antipsychotic-induced weight gain: novel preliminary data on the pharmacogenetic puzzle. J Clin Psychiatry. 2001;62 Suppl 23:45-66. PMID 11603885
- [Background] Beckers S, Zegers D, de Freitas F, Mertens IL, Van Gaal LF, Van Hul W. Association study of MC4R with complex obesity and replication of the rs17782313 association signal. Mol Genet Metab. 2011 May;103(1):71-5. doi: 10.1016/j.ymgme.2011.01.007. Epub 2011 Jan 22. PMID 21303735
- [Background] Birmaher B, Axelson D, Goldstein B, Strober M, Gill MK, Hunt J, Houck P, Ha W, Iyengar S, Kim E, Yen S, Hower H, Esposito-Smythers C, Goldstein T, Ryan N, Keller M. Four-year longitudinal course of children and adolescents with bipolar spectrum disorders: the Course and Outcome of Bipolar Youth (COBY) study. Am J Psychiatry. 2009 Jul;166(7):795-804. doi: 10.1176/appi.ajp.2009.08101569. Epub 2009 May 15. PMID 19448190
- [Background] Birmaher B, Axelson D, Strober M, Gill MK, Valeri S, Chiappetta L, Ryan N, Leonard H, Hunt J, Iyengar S, Keller M. Clinical course of children and adolescents with bipolar spectrum disorders. Arch Gen Psychiatry. 2006 Feb;63(2):175-83. doi: 10.1001/archpsyc.63.2.175. PMID 16461861
- [Background] Branson R, Potoczna N, Kral JG, Lentes KU, Hoehe MR, Horber FF. Binge eating as a major phenotype of melanocortin 4 receptor gene mutations. N Engl J Med. 2003 Mar 20;348(12):1096-103. doi: 10.1056/NEJMoa021971. PMID 12646666
- [Background] Brotons C, Ribera A, Perich RM, Abrodos D, Magana P, Pablo S, Terradas D, Fernandez F, Permanyer G. Worldwide distribution of blood lipids and lipoproteins in childhood and adolescence: a review study. Atherosclerosis. 1998 Jul;139(1):1-9. doi: 10.1016/s0021-9150(98)00056-2. PMID 9699886
- [Background] Chambers JC, Elliott P, Zabaneh D, Zhang W, Li Y, Froguel P, Balding D, Scott J, Kooner JS. Common genetic variation near MC4R is associated with waist circumference and insulin resistance. Nat Genet. 2008 Jun;40(6):716-8. doi: 10.1038/ng.156. Epub 2008 May 4. PMID 18454146
- [Background] Chen AS, Metzger JM, Trumbauer ME, Guan XM, Yu H, Frazier EG, Marsh DJ, Forrest MJ, Gopal-Truter S, Fisher J, Camacho RE, Strack AM, Mellin TN, MacIntyre DE, Chen HY, Van der Ploeg LH. Role of the melanocortin-4 receptor in metabolic rate and food intake in mice. Transgenic Res. 2000 Apr;9(2):145-54. doi: 10.1023/a:1008983615045. PMID 10951699
- [Background] Comer JS, Mojtabai R, Olfson M. National trends in the antipsychotic treatment of psychiatric outpatients with anxiety disorders. Am J Psychiatry. 2011 Oct;168(10):1057-65. doi: 10.1176/appi.ajp.2011.11010087. Epub 2011 Jul 28. PMID 21799067
- [Background] Cook S, Weitzman M, Auinger P, Nguyen M, Dietz WH. Prevalence of a metabolic syndrome phenotype in adolescents: findings from the third National Health and Nutrition Examination Survey, 1988-1994. Arch Pediatr Adolesc Med. 2003 Aug;157(8):821-7. doi: 10.1001/archpedi.157.8.821. PMID 12912790
- [Background] Correll CU, Kratochvil CJ, March JS. Developments in pediatric psychopharmacology: focus on stimulants, antidepressants, and antipsychotics. J Clin Psychiatry. 2011 May;72(5):655-70. doi: 10.4088/JCP.11r07064. PMID 21658348
- [Background] Correll CU, Lencz T, Malhotra AK. Antipsychotic drugs and obesity. Trends Mol Med. 2011 Feb;17(2):97-107. doi: 10.1016/j.molmed.2010.10.010. Epub 2010 Dec 22. PMID 21185230
- [Background] Correll CU, Malhotra AK. Pharmacogenetics of antipsychotic-induced weight gain. Psychopharmacology (Berl). 2004 Aug;174(4):477-89. doi: 10.1007/s00213-004-1949-9. Epub 2004 Jul 8. PMID 15243737
- [Background] Correll CU, Manu P, Olshanskiy V, Napolitano B, Kane JM, Malhotra AK. Cardiometabolic risk of second-generation antipsychotic medications during first-time use in children and adolescents. JAMA. 2009 Oct 28;302(16):1765-73. doi: 10.1001/jama.2009.1549. PMID 19861668
- [Background] Crystal S, Olfson M, Huang C, Pincus H, Gerhard T. Broadened use of atypical antipsychotics: safety, effectiveness, and policy challenges. Health Aff (Millwood). 2009 Sep-Oct;28(5):w770-81. doi: 10.1377/hlthaff.28.5.w770. Epub 2009 Jul 21. PMID 19622537
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] DE Hert M, Correll CU, Bobes J, Cetkovich-Bakmas M, Cohen D, Asai I, Detraux J, Gautam S, Moller HJ, Ndetei DM, Newcomer JW, Uwakwe R, Leucht S. Physical illness in patients with severe mental disorders. I. Prevalence, impact of medications and disparities in health care. World Psychiatry. 2011 Feb;10(1):52-77. doi: 10.1002/j.2051-5545.2011.tb00014.x. PMID 21379357
- [Background] De Hert M, Detraux J, van Winkel R, Yu W, Correll CU. Metabolic and cardiovascular adverse effects associated with antipsychotic drugs. Nat Rev Endocrinol. 2011 Oct 18;8(2):114-26. doi: 10.1038/nrendo.2011.156. PMID 22009159
- [Background] De Hert M, Dobbelaere M, Sheridan EM, Cohen D, Correll CU. Metabolic and endocrine adverse effects of second-generation antipsychotics in children and adolescents: A systematic review of randomized, placebo controlled trials and guidelines for clinical practice. Eur Psychiatry. 2011 Apr;26(3):144-58. doi: 10.1016/j.eurpsy.2010.09.011. Epub 2011 Feb 3. PMID 21295450
- [Background] DelBello MP, Versavel M, Ice K, Keller D, Miceli J. Tolerability of oral ziprasidone in children and adolescents with bipolar mania, schizophrenia, or schizoaffective disorder. J Child Adolesc Psychopharmacol. 2008 Oct;18(5):491-9. doi: 10.1089/cap.2008.008. PMID 18928413
- [Background] DelBello MP, Findling RL, Wang PP, Gundapaneni BP, Versavel M. Efficacy and safety of ziprasidone in pediatric bipolar disorder. Annual NCDEU Meeting, Phoenix, AZ, May 27-30, 2008.
- [Background] Dennison BA, Russo TJ, Burdick PA, Jenkins PL. An intervention to reduce television viewing by preschool children. Arch Pediatr Adolesc Med. 2004 Feb;158(2):170-6. doi: 10.1001/archpedi.158.2.170. PMID 14757609
- [Background] Dickstein DP, Towbin KE, Van Der Veen JW, Rich BA, Brotman MA, Knopf L, Onelio L, Pine DS, Leibenluft E. Randomized double-blind placebo-controlled trial of lithium in youths with severe mood dysregulation. J Child Adolesc Psychopharmacol. 2009 Feb;19(1):61-73. doi: 10.1089/cap.2008.044. PMID 19232024
- [Background] Dietz WH. Health consequences of obesity in youth: childhood predictors of adult disease. Pediatrics. 1998 Mar;101(3 Pt 2):518-25. PMID 12224658
- [Background] Findling RL, Cavus I, Pappadopulos E, Bachinsly M, Schwartz J, Vanderburg D. Efficacy and safety of ziprasidone in adolescents with schizophrenia. Presented at the 2nd Bi-annual Meeting of the Schizophrenia International Research Society (SIRS), April 10-14, 2010, Venice, Italy.
- [Background] Gibbons RD, Hedeker D, Elkin I, Waternaux C, Kraemer HC, Greenhouse JB, Shea MT, Imber SD, Sotsky SM, Watkins JT. Some conceptual and statistical issues in analysis of longitudinal psychiatric data. Application to the NIMH treatment of Depression Collaborative Research Program dataset. Arch Gen Psychiatry. 1993 Sep;50(9):739-50. doi: 10.1001/archpsyc.1993.01820210073009. PMID 8357299
- [Background] Guo SS, Roche AF, Chumlea WC, Gardner JD, Siervogel RM. The predictive value of childhood body mass index values for overweight at age 35 y. Am J Clin Nutr. 1994 Apr;59(4):810-9. doi: 10.1093/ajcn/59.4.810. PMID 8147324
- [Background] Guy W. ECDEU Assessment Manual for Psychopharmacology, revised, 1976 Vol DHEW Pub. No. (ADM) 76-338. Rockville, MD: National Institute of Mental Health.
- [Background] Heard-Costa NL, Zillikens MC, Monda KL, Johansson A, Harris TB, Fu M, Haritunians T, Feitosa MF, Aspelund T, Eiriksdottir G, Garcia M, Launer LJ, Smith AV, Mitchell BD, McArdle PF, Shuldiner AR, Bielinski SJ, Boerwinkle E, Brancati F, Demerath EW, Pankow JS, Arnold AM, Chen YD, Glazer NL, McKnight B, Psaty BM, Rotter JI, Amin N, Campbell H, Gyllensten U, Pattaro C, Pramstaller PP, Rudan I, Struchalin M, Vitart V, Gao X, Kraja A, Province MA, Zhang Q, Atwood LD, Dupuis J, Hirschhorn JN, Jaquish CE, O'Donnell CJ, Vasan RS, White CC, Aulchenko YS, Estrada K, Hofman A, Rivadeneira F, Uitterlinden AG, Witteman JC, Oostra BA, Kaplan RC, Gudnason V, O'Connell JR, Borecki IB, van Duijn CM, Cupples LA, Fox CS, North KE. NRXN3 Is a Novel Locus for Waist Circumference: A Genome-Wide Association Study from the CHARGE Consortium PLoS Genet 2009; 5: e1000539.
- [Background] Henderson DC, Cagliero E, Gray C, Nasrallah RA, Hayden DL, Schoenfeld DA, Goff DC. Clozapine, diabetes mellitus, weight gain, and lipid abnormalities: A five-year naturalistic study. Am J Psychiatry. 2000 Jun;157(6):975-81. doi: 10.1176/appi.ajp.157.6.975. PMID 10831479
- [Background] Hughes CW, Rintelmann J, Emslie GJ, Lopez M, MacCabe N. A revised anchored version of the BPRS-C for childhood psychiatric disorders. J Child Adolesc Psychopharmacol. 2001 Spring;11(1):77-93. doi: 10.1089/104454601750143500. PMID 11322749
- [Background] Huszar D, Lynch CA, Fairchild-Huntress V, Dunmore JH, Fang Q, Berkemeier LR, Gu W, Kesterson RA, Boston BA, Cone RD, Smith FJ, Campfield LA, Burn P, Lee F. Targeted disruption of the melanocortin-4 receptor results in obesity in mice. Cell. 1997 Jan 10;88(1):131-41. doi: 10.1016/s0092-8674(00)81865-6. PMID 9019399
- [Background] Kahn RS, Fleischhacker WW, Boter H, Davidson M, Vergouwe Y, Keet IP, Gheorghe MD, Rybakowski JK, Galderisi S, Libiger J, Hummer M, Dollfus S, Lopez-Ibor JJ, Hranov LG, Gaebel W, Peuskens J, Lindefors N, Riecher-Rossler A, Grobbee DE; EUFEST study group. Effectiveness of antipsychotic drugs in first-episode schizophrenia and schizophreniform disorder: an open randomised clinical trial. Lancet. 2008 Mar 29;371(9618):1085-97. doi: 10.1016/S0140-6736(08)60486-9. PMID 18374841
- [Background] Kang SJ, Chiang CW, Palmer CD, Tayo BO, Lettre G, Butler JL, Hackett R, Adeyemo AA, Guiducci C, Berzins I, Nguyen TT, Feng T, Luke A, Shriner D, Ardlie K, Rotimi C, Wilks R, Forrester T, McKenzie CA, Lyon HN, Cooper RS, Zhu X, Hirschhorn JN. Genome-wide association of anthropometric traits in African- and African-derived populations. Hum Mol Genet. 2010 Jul 1;19(13):2725-38. doi: 10.1093/hmg/ddq154. Epub 2010 Apr 16. PMID 20400458
- [Background] Katz A, Nambi SS, Mather K, Baron AD, Follmann DA, Sullivan G, Quon MJ. Quantitative insulin sensitivity check index: a simple, accurate method for assessing insulin sensitivity in humans. J Clin Endocrinol Metab. 2000 Jul;85(7):2402-10. doi: 10.1210/jcem.85.7.6661. PMID 10902785
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Kiess W, Reich A, Muller G, Meyer K, Galler A, Bennek J, Kratzsch J. Clinical aspects of obesity in childhood and adolescence--diagnosis, treatment and prevention. Int J Obes Relat Metab Disord. 2001 May;25 Suppl 1:S75-9. doi: 10.1038/sj.ijo.0801704. PMID 11466594
- [Background] Kolotkin RL, Crosby RD, Corey-Lisle PK, Li H, Swanson JM. Performance of a weight-related measure of Quality of Life in a psychiatric sample. Qual Life Res. 2006 May;15(4):587-96. doi: 10.1007/s11136-005-4627-4. PMID 16688492
- [Background] Kolotkin RL, Zeller M, Modi AC, Samsa GP, Quinlan NP, Yanovski JA, Bell SK, Maahs DM, de Serna DG, Roehrig HR. Assessing weight-related quality of life in adolescents. Obesity (Silver Spring). 2006 Mar;14(3):448-57. doi: 10.1038/oby.2006.59. PMID 16648616
- [Background] Koponen H, Saari K, Savolainen M, Isohanni M. Weight gain and glucose and lipid metabolism disturbances during antipsychotic medication: a review. Eur Arch Psychiatry Clin Neurosci. 2002 Dec;252(6):294-8. doi: 10.1007/s00406-002-0394-1. PMID 12563538
- [Background] Isolan L, Pheula G, Salum GA Jr, Oswald S, Rohde LA, Manfro GG. An open-label trial of escitalopram in children and adolescents with social anxiety disorder. J Child Adolesc Psychopharmacol. 2007 Dec;17(6):751-60. doi: 10.1089/cap.2007.0007. PMID 18315447
- [Background] Leibenluft E, Charney DS, Towbin KE, Bhangoo RK, Pine DS. Defining clinical phenotypes of juvenile mania. Am J Psychiatry. 2003 Mar;160(3):430-7. doi: 10.1176/appi.ajp.160.3.430. PMID 12611821
- [Background] Leibenluft E. Severe mood dysregulation, irritability, and the diagnostic boundaries of bipolar disorder in youths. Am J Psychiatry. 2011 Feb;168(2):129-42. doi: 10.1176/appi.ajp.2010.10050766. Epub 2010 Dec 1. PMID 21123313
- [Background] Lencz T, Lambert C, DeRosse P, Burdick KE, Morgan TV, Kane JM, Kucherlapati R, Malhotra AK. Runs of homozygosity reveal highly penetrant recessive loci in schizophrenia. Proc Natl Acad Sci U S A. 2007 Dec 11;104(50):19942-7. doi: 10.1073/pnas.0710021104. Epub 2007 Dec 5. PMID 18077426
- [Background] Lencz T, Malhotra AK. Pharmacogenetics of antipsychotic-induced side effects. Dialogues Clin Neurosci. 2009;11(4):405-15. doi: 10.31887/DCNS.2009.11.4/tlencz. PMID 20135898
- [Background] Lencz T, Morgan TV, Athanasiou M, Dain B, Reed CR, Kane JM, Kucherlapati R, Malhotra AK. Converging evidence for a pseudoautosomal cytokine receptor gene locus in schizophrenia. Mol Psychiatry. 2007 Jun;12(6):572-80. doi: 10.1038/sj.mp.4001983. Epub 2007 Mar 20. PMID 17522711
- [Background] Lieberman JA, Stroup TS, McEvoy JP, Swartz MS, Rosenheck RA, Perkins DO, Keefe RS, Davis SM, Davis CE, Lebowitz BD, Severe J, Hsiao JK; Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) Investigators. Effectiveness of antipsychotic drugs in patients with chronic schizophrenia. N Engl J Med. 2005 Sep 22;353(12):1209-23. doi: 10.1056/NEJMoa051688. Epub 2005 Sep 19. PMID 16172203
- [Background] Liebzeit KA, Markowitz JS, Caley CF. New onset diabetes and atypical antipsychotics. Eur Neuropsychopharmacol. 2001 Feb;11(1):25-32. doi: 10.1016/s0924-977x(00)00127-9. PMID 11226809
- [Background] Little, R. & Rubin D. 2002. Statistical analysis with missing data. New York, John Wiley & Sons, Inc.
- [Background] Loos RJ, Lindgren CM, Li S, Wheeler E, Zhao JH, Prokopenko I, Inouye M, Freathy RM, Attwood AP, Beckmann JS, Berndt SI; Prostate, Lung, Colorectal, and Ovarian (PLCO) Cancer Screening Trial; Jacobs KB, Chanock SJ, Hayes RB, Bergmann S, Bennett AJ, Bingham SA, Bochud M, Brown M, Cauchi S, Connell JM, Cooper C, Smith GD, Day I, Dina C, De S, Dermitzakis ET, Doney AS, Elliott KS, Elliott P, Evans DM, Sadaf Farooqi I, Froguel P, Ghori J, Groves CJ, Gwilliam R, Hadley D, Hall AS, Hattersley AT, Hebebrand J, Heid IM; KORA; Lamina C, Gieger C, Illig T, Meitinger T, Wichmann HE, Herrera B, Hinney A, Hunt SE, Jarvelin MR, Johnson T, Jolley JD, Karpe F, Keniry A, Khaw KT, Luben RN, Mangino M, Marchini J, McArdle WL, McGinnis R, Meyre D, Munroe PB, Morris AD, Ness AR, Neville MJ, Nica AC, Ong KK, O'Rahilly S, Owen KR, Palmer CN, Papadakis K, Potter S, Pouta A, Qi L; Nurses' Health Study; Randall JC, Rayner NW, Ring SM, Sandhu MS, Scherag A, Sims MA, Song K, Soranzo N, Speliotes EK; Diabetes Genetics Initiative; Syddall HE, Teichmann SA, Timpson NJ, Tobias JH, Uda M; SardiNIA Study; Vogel CI, Wallace C, Waterworth DM, Weedon MN; Wellcome Trust Case Control Consortium; Willer CJ; FUSION; Wraight, Yuan X, Zeggini E, Hirschhorn JN, Strachan DP, Ouwehand WH, Caulfield MJ, Samani NJ, Frayling TM, Vollenweider P, Waeber G, Mooser V, Deloukas P, McCarthy MI, Wareham NJ, Barroso I, Jacobs KB, Chanock SJ, Hayes RB, Lamina C, Gieger C, Illig T, Meitinger T, Wichmann HE, Kraft P, Hankinson SE, Hunter DJ, Hu FB, Lyon HN, Voight BF, Ridderstrale M, Groop L, Scheet P, Sanna S, Abecasis GR, Albai G, Nagaraja R, Schlessinger D, Jackson AU, Tuomilehto J, Collins FS, Boehnke M, Mohlke KL. Common variants near MC4R are associated with fat mass, weight and risk of obesity. Nat Genet. 2008 Jun;40(6):768-75. doi: 10.1038/ng.140. Epub 2008 May 4. PMID 18454148
- [Background] Malhotra AK, Correll CU, Chowdhury NI, Muller DJ, Gregersen PK, Lee AT, Tiwari AK, Kane JM, Fleischhacker WW, Kahn RS, Ophoff RA, Meltzer HY, Lencz T, Kennedy JL. Association between common variants near the melanocortin 4 receptor gene and severe antipsychotic drug-induced weight gain. Arch Gen Psychiatry. 2012 Sep;69(9):904-12. doi: 10.1001/archgenpsychiatry.2012.191. PMID 22566560
- [Background] Malone RP, Delaney MA, Hyman SB, Cater JR. Ziprasidone in adolescents with autism: an open-label pilot study. J Child Adolesc Psychopharmacol. 2007 Dec;17(6):779-90. doi: 10.1089/cap.2006.0126. PMID 18315450
- [Background] Marshall WA, Tanner JM. Variations in pattern of pubertal changes in girls. Arch Dis Child. 1969 Jun;44(235):291-303. doi: 10.1136/adc.44.235.291. No abstract available. PMID 5785179
- [Background] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Maayan L, Correll CU. Weight gain and metabolic risks associated with antipsychotic medications in children and adolescents. J Child Adolesc Psychopharmacol. 2011 Dec;21(6):517-35. doi: 10.1089/cap.2011.0015. Epub 2011 Dec 13. PMID 22166172
- [Background] Mundt JC, Greist JH, Gelenberg AJ, Katzelnick DJ, Jefferson JW, Modell JG. Feasibility and validation of a computer-automated Columbia-Suicide Severity Rating Scale using interactive voice response technology. J Psychiatr Res. 2010 Dec;44(16):1224-8. doi: 10.1016/j.jpsychires.2010.04.025. Epub 2010 Jun 2. PMID 20553851
- [Background] Must A, Jacques PF, Dallal GE, Bajema CJ, Dietz WH. Long-term morbidity and mortality of overweight adolescents. A follow-up of the Harvard Growth Study of 1922 to 1935. N Engl J Med. 1992 Nov 5;327(19):1350-5. doi: 10.1056/NEJM199211053271904. PMID 1406836
- [Background] Okasora K, Takaya R, Tokuda M, Fukunaga Y, Oguni T, Tanaka H, Konishi K, Tamai H. Comparison of bioelectrical impedance analysis and dual energy X-ray absorptiometry for assessment of body composition in children. Pediatr Int. 1999 Apr;41(2):121-5. doi: 10.1046/j.1442-200x.1999.4121048.x. PMID 10221012
- [Background] Olfson M, Blanco C, Liu L, Moreno C, Laje G. National trends in the outpatient treatment of children and adolescents with antipsychotic drugs. Arch Gen Psychiatry. 2006 Jun;63(6):679-85. doi: 10.1001/archpsyc.63.6.679. PMID 16754841
- [Background] Olfson M, Crystal S, Huang C, Gerhard T. Trends in antipsychotic drug use by very young, privately insured children. J Am Acad Child Adolesc Psychiatry. 2010 Jan;49(1):13-23. doi: 10.1097/00004583-201001000-00005. PMID 20215922
- [Background] Pandina GJ, Aman MG, Findling RL. Risperidone in the management of disruptive behavior disorders. J Child Adolesc Psychopharmacol. 2006 Aug;16(4):379-92. doi: 10.1089/cap.2006.16.379. PMID 16958564
- [Background] Parsons B, Allison DB, Loebel A, Williams K, Giller E, Romano S, Siu C. Weight effects associated with antipsychotics: a comprehensive database analysis. Schizophr Res. 2009 May;110(1-3):103-10. doi: 10.1016/j.schres.2008.09.025. Epub 2009 Mar 24. PMID 19321312
- [Background] Price AL, Patterson NJ, Plenge RM, Weinblatt ME, Shadick NA, Reich D. Principal components analysis corrects for stratification in genome-wide association studies. Nat Genet. 2006 Aug;38(8):904-9. doi: 10.1038/ng1847. Epub 2006 Jul 23. PMID 16862161
- [Background] Psychological Corporation (1999): Wechsler Abbreviated Scale of Intelligence (WASI) manual. San-Antonio, Tx.
- [Background] Qi L, Kraft P, Hunter DJ, Hu FB. The common obesity variant near MC4R gene is associated with higher intakes of total energy and dietary fat, weight change and diabetes risk in women. Hum Mol Genet. 2008 Nov 15;17(22):3502-8. doi: 10.1093/hmg/ddn242. Epub 2008 Aug 12. PMID 18697794
- [Background] Raper N, Perloff B, Ingwersen L, Steinfeldt L, Anand J. An overview of USDA's dietary intake data system. Journal of Food Composition and Analysis 2004; 17;545-55.
- [Background] Ridker PM. C-reactive protein, inflammation, and cardiovascular disease: clinical update. Tex Heart Inst J. 2005;32(3):384-6. No abstract available. PMID 16392225
- [Background] Rifai N, Warnick GR, McNamara JR, Belcher JD, Grinstead GF, Frantz ID Jr. Measurement of low-density-lipoprotein cholesterol in serum: a status report. Clin Chem. 1992 Jan;38(1):150-60. PMID 1733589
- [Background] Robinson DG, Woerner MG, Napolitano B, Patel RC, Sevy SM, Gunduz-Bruce H, Soto-Perello JM, Mendelowitz A, Khadivi A, Miller R, McCormack J, Lorell BS, Lesser ML, Schooler NR, Kane JM. Randomized comparison of olanzapine versus risperidone for the treatment of first-episode schizophrenia: 4-month outcomes. Am J Psychiatry. 2006 Dec;163(12):2096-102. doi: 10.1176/ajp.2006.163.12.2096. PMID 17151160
- [Background] Rosenfeld JA, Malhotra AK, Lencz T. Novel multi-nucleotide polymorphisms in the human genome characterized by whole genome and exome sequencing. Nucleic Acids Res. 2010 Oct;38(18):6102-11. doi: 10.1093/nar/gkq408. Epub 2010 May 20. PMID 20488869
- [Background] Safer DJ. A comparison of risperidone-induced weight gain across the age span. J Clin Psychopharmacol. 2004 Aug;24(4):429-36. doi: 10.1097/01.jcp.0000130558.86125.5b. PMID 15232335
- [Background] Scherag A, Jarick I, Grothe J, Biebermann H, Scherag S, Volckmar AL, Vogel CI, Greene B, Hebebrand J, Hinney A. Investigation of a genome wide association signal for obesity: synthetic association and haplotype analyses at the melanocortin 4 receptor gene locus. PLoS One. 2010 Nov 15;5(11):e13967. doi: 10.1371/journal.pone.0013967. PMID 21085626
- [Background] Sikich L, Frazier JA, McClellan J, Findling RL, Vitiello B, Ritz L, Ambler D, Puglia M, Maloney AE, Michael E, De Jong S, Slifka K, Noyes N, Hlastala S, Pierson L, McNamara NK, Delporto-Bedoya D, Anderson R, Hamer RM, Lieberman JA. Double-blind comparison of first- and second-generation antipsychotics in early-onset schizophrenia and schizo-affective disorder: findings from the treatment of early-onset schizophrenia spectrum disorders (TEOSS) study. Am J Psychiatry. 2008 Nov;165(11):1420-31. doi: 10.1176/appi.ajp.2008.08050756. Epub 2008 Sep 15. PMID 18794207
- [Background] Snitker S, Le KY, Hager E, Caballero B, Black MM. Association of physical activity and body composition with insulin sensitivity in a community sample of adolescents. Arch Pediatr Adolesc Med. 2007 Jul;161(7):677-83. doi: 10.1001/archpedi.161.7.677. PMID 17606831
- [Background] Simpson GM, Angus JW. A rating scale for extrapyramidal side effects. Acta Psychiatr Scand Suppl. 1970;212:11-9. doi: 10.1111/j.1600-0447.1970.tb02066.x. No abstract available. PMID 4917967
- [Background] Strom BL, Eng SM, Faich G, Reynolds RF, D'Agostino RB, Ruskin J, Kane JM. Comparative mortality associated with ziprasidone and olanzapine in real-world use among 18,154 patients with schizophrenia: The Ziprasidone Observational Study of Cardiac Outcomes (ZODIAC). Am J Psychiatry. 2011 Feb;168(2):193-201. doi: 10.1176/appi.ajp.2010.08040484. Epub 2010 Nov 1. PMID 21041245
- [Background] Stutzmann F, Cauchi S, Durand E, Calvacanti-Proenca C, Pigeyre M, Hartikainen AL, Sovio U, Tichet J, Marre M, Weill J, Balkau B, Potoczna N, Laitinen J, Elliott P, Jarvelin MR, Horber F, Meyre D, Froguel P. Common genetic variation near MC4R is associated with eating behaviour patterns in European populations. Int J Obes (Lond). 2009 Mar;33(3):373-8. doi: 10.1038/ijo.2008.279. Epub 2009 Jan 20. PMID 19153581
- [Background] Tyrrell VJ, Richards G, Hofman P, Gillies GF, Robinson E, Cutfield WS. Foot-to-foot bioelectrical impedance analysis: a valuable tool for the measurement of body composition in children. Int J Obes Relat Metab Disord. 2001 Feb;25(2):273-8. doi: 10.1038/sj.ijo.0801531. PMID 11410831
- [Background] Tanner JM, Whitehouse RH. Clinical longitudinal standards for height, weight, height velocity, weight velocity, and stages of puberty. Arch Dis Child. 1976 Mar;51(3):170-9. doi: 10.1136/adc.51.3.170. PMID 952550
- [Background] Tiwari AK, Zai CC, Likhodi O, Lisker A, Singh D, Souza RP, Batra P, Zaidi SH, Chen S, Liu F, Puls I, Meltzer HY, Lieberman JA, Kennedy JL, Muller DJ. A common polymorphism in the cannabinoid receptor 1 (CNR1) gene is associated with antipsychotic-induced weight gain in Schizophrenia. Neuropsychopharmacology. 2010 May;35(6):1315-24. doi: 10.1038/npp.2009.235. Epub 2010 Jan 27. PMID 20107430
- [Background] Valladares M, Dominguez-Vasquez P, Obregon AM, Weisstaub G, Burrows R, Maiz A, Santos JL. Melanocortin-4 receptor gene variants in Chilean families: association with childhood obesity and eating behavior. Nutr Neurosci. 2010 Apr;13(2):71-8. doi: 10.1179/147683010X12611460763643. PMID 20406574
- [Background] Vanhala M. Childhood weight and metabolic syndrome in adults. Ann Med. 1999 Aug;31(4):236-9. doi: 10.3109/07853899908995885. PMID 10480753
- [Background] Waxmonsky J, Pelham WE, Gnagy E, Cummings MR, O'Connor B, Majumdar A, Verley J, Hoffman MT, Massetti GA, Burrows-MacLean L, Fabiano GA, Waschbusch DA, Chacko A, Arnold FW, Walker KS, Garefino AC, Robb JA. The efficacy and tolerability of methylphenidate and behavior modification in children with attention-deficit/hyperactivity disorder and severe mood dysregulation. J Child Adolesc Psychopharmacol. 2008 Dec;18(6):573-88. doi: 10.1089/cap.2008.065. PMID 19108662
- [Background] Wu L, Xi B, Zhang M, Shen Y, Zhao X, Cheng H, Hou D, Sun D, Ott J, Wang X, Mi J. Associations of six single nucleotide polymorphisms in obesity-related genes with BMI and risk of obesity in Chinese children. Diabetes. 2010 Dec;59(12):3085-9. doi: 10.2337/db10-0273. Epub 2010 Sep 15. PMID 20843981

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 subjects were consented to the study and received screening, 7 subjects did not meet the eligibility criteria to the study and were therefore not randomized to the study
Groups:
- Ziprasidone: (20-160mg/d, bid) for 12 weeks
  Ziprasidone: random assignment to ZIP (20-160mg/d, bid dosing)
  4 participants
- Aripiprazole, Quetiapine, Risperidone: Aripiprazole (2-30mg/d), Quetiapine (25-800mg/d) or Risperidone (0.1-8mg/d) for 12 weeks
  aripiprazole, quetiapine, or risperidone: random assignement to Usual Care antipsychotic UC antipsychotic (aripiprazole 2-30mg/d, quetiapine 25-800mg/d or risperidone 0.1-8mg/d)
  3 participants
Period: Overall Study
Arm/Group | Ziprasidone | Aripiprazole, Quetiapine, Risperidone
Started | 4 | 3
Completed | 1 | 2
Not Completed | 3 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — refused medication switch | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — stopped taking meds | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ziprasidone: (20-160mg/d, bid) for 12 weeks
  Ziprasidone: random assignment to ZIP (20-160mg/d, bid dosing)
  4 patients were randomized to Ziprasidone
- Aripiprazole, Quetiapine, Risperidone: Aripiprazole (2-30mg/d), Quetiapine (25-800mg/d) or Risperidone (0.1-8mg/d) for 12 weeks
  aripiprazole, quetiapine, or risperidone: random assignement to Usual Care antipsychotic UC antipsychotic (aripiprazole 2-30mg/d, quetiapine 25-800mg/d or risperidone 0.1-8mg/d)
  3 patients were randomized to usual care
- Total: Total of all reporting groups
Arm/Group | Ziprasidone | Aripiprazole, Quetiapine, Risperidone | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Time Frame: baseline to week 12
Measure: Mean (Standard Deviation); unit: lbs
Groups:
- Ziprasidone: (20-160mg/d, bid) for 12 weeks
  Ziprasidone: random assignment to ZIP (20-160mg/d, bid dosing)
  4 participants, only one completed study and he was questionable compliant, no sufficient data for weight changes
- Aripiprazole, Quetiapine, Risperidone: Aripiprazole (2-30mg/d), Quetiapine (25-800mg/d) or Risperidone (0.1-8mg/d) for 12 weeks
  aripiprazole, quetiapine, or risperidone: random assignement to Usual Care antipsychotic UC antipsychotic (aripiprazole 2-30mg/d, quetiapine 25-800mg/d or risperidone 0.1-8mg/d)
  3 participants, only two completed study, no sufficient data for weight changes
Arm/Group | Ziprasidone | Aripiprazole, Quetiapine, Risperidone
Number analyzed (Participants) | 4 | 3
lbs
  baseline | 120.5 (8.23) | 118.5 (27.92)
  week 12 (n=1,2) | 151 (0) | 141 (7.06)

2. Secondary Outcome: Percent Weight Change Compared to Baseline Weight
Time Frame: baseline to week 12
Measure: Mean (Standard Deviation); unit: percentage of weight change
Arm/Group | Ziprasidone | Aripiprazole, Quetiapine, Risperidone
Number analyzed (Participants) | 1 | 2
percentage of weight change | 11.58 (0) | 5.66 (4.66)

3. Secondary Outcome: BMI Z-scores
Time Frame: baseline to week 12
Measure: Mean (Standard Deviation); unit: BMI z-score
Arm/Group | Ziprasidone | Aripiprazole, Quetiapine, Risperidone
Number analyzed (Participants) | 4 | 3
BMI z-score
  baseline | -0.51 (0.55) | -0.37 (1.05)
  week 12 (n=1, n=2) | 0.22 (0) | 0.38 (0.85)

4. Secondary Outcome: BMI Percentile
Time Frame: baseline to week 12
Measure: Mean (Standard Deviation); unit: BMI percentile
Arm/Group | Ziprasidone | Aripiprazole, Quetiapine, Risperidone
Number analyzed (Participants) | 4 | 3
BMI percentile
  baseline | 32 (20.31) | 37.67 (36.66)
  week 12 (n=1, n=2) | 59 (1) | 62.5 (30.41)

ADVERSE EVENTS:
Groups:
- Ziprasidone: (20-160mg/d, bid) for 12 weeks
  Ziprasidone: random assignment to ZIP (20-160mg/d, bid dosing)
  4 participants, only one completed study and he was questionable compliant, no sufficient data for weight changes
  there were no serious adverse events in this group
- Aripiprazole, Quetiapine, Risperidone: Aripiprazole (2-30mg/d), Quetiapine (25-800mg/d) or Risperidone (0.1-8mg/d) for 12 weeks
  aripiprazole, quetiapine, or risperidone: random assignement to Usual Care antipsychotic UC antipsychotic (aripiprazole 2-30mg/d, quetiapine 25-800mg/d or risperidone 0.1-8mg/d)
  3 participants, only two completed study, no sufficient data for weight changes
  there were no serious adverse events in this group
Arm/Group | Ziprasidone | Aripiprazole, Quetiapine, Risperidone
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No